CLINICAL TRIAL: NCT00576277
Title: A Prospective, Double-Blind, Randomized, Placebo-Controlled Trial of AV411 to Assess Its Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy in the Treatment of Neuropathic Pain
Brief Title: Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of AV411 in Neuropathic Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Avigen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AV411-010
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Last update posted 2007-12-19 (Estimated); Status verified 2007-04

CONDITIONS: Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — ibudilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: AV411

SUMMARY:
The purpose of this study is to determine the safety, tolerability and pharmacokinetics of AV411 after single and multiple doses in patients with chronic neuropathic pain due to diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetic neuropathy or complex regional pain syndrome of at least 6 months duration
* VAS score of 4 cm or higher at Screening
* No clinical abnormality in laboratory and urine analyses
* Electrocardiogram within normal limits at Screening
* Negative pregnancy test on Study Day 1 for female subjects of childbearing potential
* On stable doses of medications, analgesic or others for at least 8 weeks prior to study enrollment
* Willing to use barrier contraceptive during the period of the study

Exclusion Criteria:

* Known hypersensitivity to AV411 or its components
* Conditions which might affect drug absorption, metabolism or excretion
* Untreated mental illness, current drug addiction or abuse or alcoholism
* Donated blood in the past 90 days or have poor peripheral venous access
* Platelets <100,000mm3 or a history of thrombocytopenia
* Known or suspected chronic liver disease
* GFR <=90mL/min/1.73m2 (Cockcroft-Gault)
* Female subjects who are pregnant or nursing mothers
* Received an investigational drug in the past 90 days
* Unable to swallow large capsules

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2006-09; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Safety
Tolerability
Pharmacokinetic profile
Pharmacodynamic profile

SECONDARY OUTCOMES:
Brief Pain Inventory
Visual Analog Scale
Clinical Global Impression of Change
Use of analgesic or adjuvant medications for neuropathic pain
Correlation between plasma concentrations of AV411 and pain intensity assessments

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - University of Adelaide, Adelaide
  - Peninsular Specialist Centre, Kipparing